CLINICAL TRIAL: NCT00860652
Title: Radiotherapy - Adjuvant Versus Early Salvage. A Phase III Multi-centre Randomised Trial Comparing Adjuvant Radiotherapy (RT) With Early Salvage RT in Patients With Positive Margins or Extraprostatic Disease Following Radical Prostatectomy.
Brief Title: Radiotherapy - Adjuvant Versus Early Salvage
Acronym: RAVES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Urological Society of Australia and New Zealand (USANZ) (Unknown); Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 08.03
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Prostate Cancer
Keywords: Oncology; Prostate Cancer; Radiotherapy; Radical Prostatectomy; Prior Radical Prostatectomy (RP); Histological Confirmation of adenocarcinoma of the prostate; Positive margins and/or extraprostatic extension (EPE)
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Radiotherapy, Adjuvant; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant Radiotherapy (RT) (Experimental): Adjuvant Radiotherapy (64Gy in 32 Fractions to the prostate bed)
  Interventions: Radiation: Adjuvant Radiotherapy
- Active Surveillance with Early SalvageRT (Experimental): Active Surveillance with Early Salvage Radiotherapy
  Interventions: Radiation: Early Salvage Radiotherapy

INTERVENTIONS:
Radiation: Adjuvant Radiotherapy — Adjuvant RT (ART) commenced within 4 months of Radical Prostatectomy. 64Gy in 32 fractions to the prostate bed.
  Other Names: ART, Radiation
  Arms: Adjuvant Radiotherapy (RT)
Radiation: Early Salvage Radiotherapy — Active surveillance with early Salvage RT (SRT). SRT - 64Gy in 32 fractions to the prostate bed. RT should commence no later than 4 months following the first PSA measurement ≥ 0.2ng/mL.
  Other Names: SRT, Surveillance, Radiation
  Arms: Active Surveillance with Early SalvageRT

SUMMARY:
Radical prostatectomy (RP) is the most common curative approach offered to men with newly diagnosed prostate cancer. Unfortunately, up to half of these patients will have factors placing them at high risk of their cancer recurring. Having radiotherapy after RP is known to improve cure rates, but what is not known is whether it should be given straight after the operation or only when there is a rising PSA after surgery indicating active cancer. Immediate RT may not benefit all men, and can cause serious side effects such as bladder and bowel problems and impotence. International lack of consensus on the optimal timing of RT has resulted in varied clinical practice. This phase 3 trial will compare the two approaches.

DETAILED DESCRIPTION:
This is a prospective, multi-centre, international, randomised controlled trial with a 1:1 allocation ratio. Patients with positive margins and/or pT3 disease will be randomised to adjuvant RT (Standard Arm) or active surveillance with salvage RT delivered at early relapse (Experimental Arm). 64 Gy in 32 fractions will be delivered to the prostate bed. QoL self-assessment questionnaires, Hospital Anxiety and Depression Score and toxicity will be assessed at baseline, the end of RT and annually for 5 years. Patients will be seen by their doctor 6 monthly for the first 5 years, then annually for the next 5 years. A blood test measuring prostate specific antigen (PSA) is done 3 monthly for the first 5 years for patients randomised to early salvage RT, then 6 monthly from years 5 to 10.

ELIGIBILITY:
Inclusion Criteria:

* Prior Radical Prostatectomy (RP) for adenocarcinoma of the prostate.
* Histological confirmation of adenocarcinoma of the prostate with the Gleason score reported (Radical Prostatectomy specimen).
* Patients must have at least one of the following risk factors: 1) Positive margins, 2) Extraprostatic extension (EPE) with or without seminal vesicle involvement (pT3a or pT3b)
* Capable of starting RT within 4 months of RP (a requirement if randomised to adjuvant RT arm)
* Most recent PSA ≤ 0.10 ng/ml following RP and prior to randomisation
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
* Patient able to adhere to the specified follow-up schedule and complete the Quality of Life and anxiety/depression self-assessments
* Written informed consent obtained prior to randomisation
* Completion of all pre-treatment evaluations
* 18 years and older

Exclusion Criteria:

* Previous pelvic RT
* Androgen deprivation (AD) prior to or following RP
* Evidence of nodal or distant metastases
* Co-morbidities that would interfere with the completion of treatment and/or 5 years of follow-up
* Concurrent cytotoxic medication
* Hip prosthesis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2009-03-03 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Biochemical failure: PSA ≥ 0.4 ng/ml and rising following RT | After 160 events have been observed, expected to be 5 years after recruitment closes

SECONDARY OUTCOMES:
Quality of Life | Final Analysis will be after 160 events, estimated to be five years after the end of accrual
Toxicity | Final analysis will be after 160 events, estimated to be 5 years after end of accrual.
Anxiety/Depression | Final analysis will be after 160 events, estimated to be 5 years after end of accrual.
Biochemical failure-free survival | Final analysis will be after 160 events, estimated to be 5 years after end of accrual.
Overall survival | Final analysis will be after 160 events, estimated to be 5 years after end of accrual.
Disease-specific survival | Final analysis will be after 160 events, estimated to be 5 years after end of accrual.
Time to distant failure | Final analysis will be after 160 events, estimated to be 5 years after end of accrual.
Time to local failure | Final analysis will be after 160 events, estimated to be 5 years after end of accrual.
Time to the initiation of androgen ablation | Final analysis will be after 160 events, estimated to be 5 years after end of accrual.
Quality adjusted life years | Final analysis will be after 160 events, estimated to be 5 years after end of accrual.
Cost-utility | Final analysis will be after 160 events, estimated to be 5 years after end of accrual.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pearse, MBChB, Study Chair — Trans Tasman Radiation Oncology Group; Andrew Kneebone, Study Chair — Trans Tasman Radiation Oncology Group
Locations (36):
- Australia (30):
  - Campbelltown Hopsital, Campbelltown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Coffs Harbour Health Campus, NCCI, Coffs Harbour, New South Wales
  - Radiation Oncology Associates, Darlinghurst, New South Wales
  - St Vincent's Clinic, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Central West Cancer Services (Orange Health), Orange, New South Wales
  - Port Macquarie Base Hospital, NCCI, Port Macquarie, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Radiation Oncology Gold Coast, Gold Coast, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Oceania Oncology, Nambour, Queensland
  - Radiation Oncology - Mater Centre, South Brisbane, Queensland
  - Toowoomba Cancer Research Centre, Toowoomba, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Premion, Tugun, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Austin Hospital, Heidelberg West, Victoria
  - The Alfred/WBRC, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Perth Radiation Oncology, Perth, Western Australia
- New Zealand (6):
  - Auckland Radiation Oncology, Epsom, Auckland
  - Wellington Hospital, Newtown, Wellington Region
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Palmerston North Hospital, Palmerston North

REFERENCES:
- [Derived] Kneebone A, Fraser-Browne C, Duchesne GM, Fisher R, Frydenberg M, Herschtal A, Williams SG, Brown C, Delprado W, Haworth A, Joseph DJ, Martin JM, Matthews JHL, Millar JL, Sidhom M, Spry N, Tang CI, Turner S, Wiltshire KL, Woo HH, Davis ID, Lim TS, Pearse M. Adjuvant radiotherapy versus early salvage radiotherapy following radical prostatectomy (TROG 08.03/ANZUP RAVES): a randomised, controlled, phase 3, non-inferiority trial. Lancet Oncol. 2020 Oct;21(10):1331-1340. doi: 10.1016/S1470-2045(20)30456-3. PMID 33002437
- See also: Trans Tasman Radiation Oncology Group — http://www.trog.com.au